CLINICAL TRIAL: NCT05376345
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of BCMA-targeted LCAR-BCDR Cells Product in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: BCMA-targeted LCAR-BCDR Cells in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per sponsor request
Sponsor: Weijun Fu (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor-Investigator, Weijun Fu, Principal Investigator, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM2L202103
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LCAR-BCDR cells product (Experimental): Each subject will receive LCAR-BCDR cells
  Interventions: Biological: LCAR-BCDR cells product

INTERVENTIONS:
Biological: LCAR-BCDR cells product — Before treatment with LCAR-BCDR cells, subjects will receive a conditioning regimen

SUMMARY:
This is a prospective, single-arm, open-label, dose-finding and dose-expansion study that evaluates the safety, tolerability, PK, and anti-tumor efficacy of LCAR-BCDR cell preparations in relapsed/refractory multiple myeloma subjects who received adequate standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in the clinical study; Fully understand and be Informed of the study and sign the Informed consent (Informed Consent Form, ICF); Willing to follow and able to complete all test procedures; Informed consent must be obtained before initiating any tests or procedures related to the study that are not part of the standard treatment of the subject's disease;
2. Subjects ≥ 18 years of age.
3. Documented initial diagnosis of MM according to IMWG diagnostic criteria.
4. Presence of measurable disease at screening.
5. Received a PI and an IMiD (except thalidomide).
6. Received at least 3 prior lines of therapy for multiple myeloma, undergone at least 1 complete cycle of treatment for each line, unless progressive disease (PD) was documented by IMWG criteria as the best response to the regimen. Also, subjects refractory or intolerant to any PI and any IMiD in their previous treatment afterwards are eligible.
7. Expected survival ≥ 3 months.
8. Clinical laboratory values meet screening visit criteria
9. Fertile women must be negative using a highly sensitive serum pregnancy test (β human chorionic gonadotropin [β -HCG]) at screening time and before initial treatment with cyclophosphamide and fludarabine;

Exclusion Criteria:

1. No response to prior BCMA-targeted CAR-T therapy (except in subjects who relapsed after CR to prior CAR-T treatment).
2. Prior treatment with any antibody targeting BCMA.
3. Diagnosed or pretreated for an invasive malignancy other than multiple myeloma.
4. Prior anti-tumor treatment (before pretreatment) with insufficient washout period.
5. Known active, or prior history of central nervous system (CNS) involvement, or clinical signs of membrane/spinal membrane involvement of multiple myeloma.
6. Positive of any hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), human immunodeficiency virus antibody (HIV-Ab) at the time of screening.
7. Serious underlying medical conditions
8. Male subjects who have a birth plan during the study period or within 1 year after the study treatment.
9. Female subjects who are pregnant, breast-feeding, or plan to become pregnant during the study period or within 1 year after the study treatment.
10. The investigator considered that the subjects were not suitable for any conditions of participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Recommended Phase 2 dose (RP2D) finding | 30 days after LCAR-BCDR infusion (Day 1)
  RP2D established through ATD+BOIN design
CAR positive T cells in peripheral blood and bone marrow | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  CAR positive T cells in peripheral blood and bone marrow after LCAR-BCDR infusion
CAR transgene levels in peripheral blood and bone marrow | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  CAR transgene levels in peripheral blood and bone marrow after LCAR-BCDR infusion

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  The ORR is defined as the percentage of participants who achieve partial response (PR) or better according to international myeloma working group (IMWG) criteria.
Progression-free survival (PFS) | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LCAR-BCDR to the first documented disease progression (according to IMWG criteria) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-AIO to death of the subject
Incidence of anti-LCAR-BCDR antibody | Minimum 2 years after LCAR-BCDR infusion (Day 1)
  Venous blood samples will be collected to measure LCAR-BCDR positive cell concentrations and the transgenic level of LCAR-BCDR, at the time points when anti-LCAR-BCDR antibody serum samples are evaluated

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Gobroad Boren Hospital, Beijing, Beijing Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Fourth People's Hospital Affiliated to Tongji University, Shanghai
  - Institute of Hematology & Blood Diseases Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou

IPD SHARING:
Plan to Share IPD: No